CLINICAL TRIAL: NCT05427513
Title: Efficacy of Tranexamic Acid in Preventing Post Operative Blood Loss and Associated Complications in Bone Sarcoma Patients Treated With Limb Salvage Surgery: A Randomized Controlled Trial
Brief Title: Efficacy of Tranexamic Acid in Preventing Post Operative Blood Loss in Bone Sarcoma Patient
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-22-07
Record Dates: First submitted 2022-04-06; First posted 2022-06-22 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): will injection 10 ml of normal saline to ensure binding
  Interventions: Other: normal saline
- tranexamic acid(TXA) (Active Comparator): will inject tranexamic acid according to body weight
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — will inject tranexamic acid in limb salvage surgery of sarcoma patient to check its efficacy in preventing blood loss
  Arms: tranexamic acid(TXA)
Other: normal saline — normal saline will be injected to ensure placebo
  Arms: placebo

SUMMARY:
investigator will see the efficacy of tranexamic acid in limb salvage surgery patients which will prevent blood loss and help in conservation of blood products.

ELIGIBILITY:
Inclusion Criteria:

* Limb sarcoma of upper and lower limb
* Limb salvage

Exclusion Criteria:

* liver insufficiency
* renal insufficiency
* allergic to drug
* history of thromboembolic condition
* pregnancy
* metastatic disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
blood loss | 72 hour post operatively
  measure by hemoglobin direct method
no of blood transfused | 72 hour
  measured by number of transfusion

SECONDARY OUTCOMES:
duration of hospital stay | total hospital stay post operatively for 02 month
  Total days of hospital admission 2 months after surgery
volume of drain out put | measure till drain out in 72 hour
  to measure blood collected in drain bottle
thromboembolic events | observed for 6 week determine on out patient visits
  look for limb swelling for deep vein thrombosis and chest symptoms for any embolic event confirmed by CT chest

CONTACTS AND LOCATIONS:
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital & Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
will start recruiting patient of bone sarcoma in two groups having double blinded & tranexamic acid efficacy will be checked

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT05427513/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT05427513/ICF_001.pdf